CLINICAL TRIAL: NCT02991326
Title: Osteopathic Manipulative Treatment Effect in Individuals With Temporomandibular Disorder Who Make Use of Occlusal Splints
Brief Title: Osteopathic Manipulative Treatment in Individuals With Temporomandibular Disorder Who Make Use of Occlusal Splints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Simone Saldanha Oliveira, Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Simone Oliveira
Record Dates: First submitted 2016-12-07; First posted 2016-12-13 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Temporomandibular Disorder
Keywords: Osteopathic Manipulative Treatment; Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Group (TG) (Experimental): The Individuals who already is subject to Clinical Treatment with splints offered at the Occlusion Clinic will be subject to Osteopathic Manipulative Treatment - OMT.
  Interventions: Other: Osteopathic Manipulative Treatment
- Control Group (CG) (Sham Comparator): The Individuals who already is subject to Clinical Treatment with splints offered at the Occlusion Clinic will be subject to sham intervention (Osteopathic Manipulative Treatment simulated).
  Interventions: Other: Sham intervention

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment — The Osteopathic manipulative treatment will follow the approach bellow (using latex gloves for intra oral techniques):
  * Compression of the fourth ventricle;
  * inhibitory intra-oral pressure technique (IPT) of the temporal muscle;
  * inhibition of the inferior head of the lateral pterygoid muscle;
  * intra-oral inhibition of the masseter muscle;
  * Balanced ligamentous tension (BLT) of the accessory ligaments - sphenopalatine;
  * BLT of the accessory ligaments - pterygomandibular raphe;
  * sphenopalatine ganglion technique;
  * Craniosacral rebalancing;
  Arms: Test Group (TG)
Other: Sham intervention — The sham intervention will be made in the same examination table and the same position, with the use of the latex gloves, to simulate the Osteopathic Manipulative Treatment, only doing simple touches without therapeutic effect intention.
  Arms: Control Group (CG)

SUMMARY:
This study aim to contribute with the investigation of the therapeutic effect of osteopathic manipulative treatment in pain intensity and Quality of Life in individuals diagnosed with temporomandibular disorder who make use of occlusal splints.

DETAILED DESCRIPTION:
Objective:

It is known the multifactorial etiology of Temporomandibular Disorders(TMD) which raises the need of a multidisciplinary approach for its treatment. Studies have presented good results about the use of occlusal splints along with other therapies. The Osteopathic Manipulative Treatment(OMT) has as characteristic the philosophy of global approach and precise functional diagnosis. Based on a lack of randomized blind trials about this subject, This study aim to contribute with the investigation of the therapeutic effect OMT in pain intensity and Quality of Life in participants diagnosed with TMD making use of occlusal splints.

Methodology:

This study is a randomized blind trial, with sample composed by 18 participants referred to the occlusion clinic of Fluminense Federal University (UFF), diagnosed by the team of dentists and interns of occlusion clinic through the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD). The participants will complete the Short Form 36 Health Survey(SF-36) to measure the quality of life, and pain intensity diagram with Numeric Rating Scale (NRS) to measure the pain intensity. The sample will be randomized into 2 groups (9 individuals for each): Test Group (TG) - patients subject to Clinical Treatment with splints (CT) offered at the Occlusion Clinic unit along with Osteopathic Manipulative Treatment - OMT. Control Group (CG) - patients subject only to CT and will receive a sham treatment that simulate the OMT to blind these participants. After the treatment, patients will be re-evaluated in 8 weeks' time.

Statistical analysis:

The SF-36 and the pain intensity and the most intense pain evaluation diagram with Numeric Rating Scale (NRS) will be performed by the Wilcoxon's non parametric test.

ELIGIBILITY:
Inclusion Criteria:

* individuals who has diagnosis of Temporomandibular disorder.

Exclusion Criteria:

* individuals who already has subjected to osteopathic manipulative treatment to temporomandibular disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change from Numeric Rating Scale (NRS) to measure the pain intensity at 2 month | 2 months
  The use of Numeric Rating Scale (NRS) to measure the pain intensity in each body area related by the individuals before and 2 months after the first intervention.

SECONDARY OUTCOMES:
Change from Numeric Rating Scale (NRS) for the body area with the Worst Pain(WP) at 2 months | 2 months
  The use of Numeric Rating Scale (NRS) to measure de pain intensity in the body area with the most intensity pain related by the individuals before and 2 months after first intervention.
Change from Quality of Life Survey by Short Form 36 Health Survey(SF-36) at 2 months | 2 months
  The use of SF36 to measure the score of quality of life before and 2 months after first intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe RT Goulart, Graduated, Principal Investigator — Federal Fluminense University
Locations (1):
- Federal Fuminense University, Niterói, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided